CLINICAL TRIAL: NCT05949450
Title: Prognostic Role of Troponin Dosed at 3 to 6 Months in the Evolution of Acute Myocarditis
Brief Title: Prognostic Role of High Sensitivity Troponin During Follow up in the Evolution of Acute Myocarditis
Acronym: PROGNOSTIC
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC23.0091; 2023-A0078-37 (Other: IDRCB)
Record Dates: First submitted 2023-06-08; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-06

CONDITIONS: Myocarditis
Keywords: myocarditis; troponine us
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to observe if ultra-sensitive troponins (us) measurement between 3 and 6 months after the acute event will be sensitive enough to dispense with all other examinations, particularly cardiac magnetic resonance imaging (MRI), in patients suffering from myocarditis.

The investigators will collect patient events by telephone, once a year for 4 years.

DETAILED DESCRIPTION:
Myocarditis is a frequent pathology with a heterogeneous initial clinical presentation. The long-term course of the disease is variable, with the possibility of healing and recovery, but also the likelihood of long-term deterioration, with the development of true dilated cardiomyopathy. While diagnostic criteria in the initial phase are well codified, notably with cardiac MRI, follow-up methods are less standardized. Re-evaluation between 3 and 6 months is not carried out by all teams, and if it is, the examinations performed vary from one team to another. Grenoble team has demonstrated the prognostic role of MRI reassessment at 3 and 6 months. It is also common to measure troponins to detect chronic myocarditis. However, this assay has evolved over time with the advent of ultra-sensitive troponins (us). These appear to be much more sensitive, and this increased sensitivity may lead to a change in care strategies.

For example, in the management of chest pain in emergency departments before the era of us troponins, the use of coronary CT scans improved patient management. This benefit of imaging has disappeared since the advent of troponin us.

The hypothesis of investigators is that troponin us measurement between 3 and 6 months after the acute event will be sensitive enough to dispense with all other examinations, particularly cardiac MRI, in order to identify patients at risk of poor prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients over 18 years of age
* Patients hospitalized at Grenoble Alpes University Hospital and Lyon University Hospital between June 2016 and June 2025
* Having presented chest pain and ≥1 diagnostic criteria or if no chest pain, presence of ≥2 diagnostic criteria below :

  * Electrical abnormalities (supra- or sub-ST, T-wave inversion, atrioventricular blocks 1-3 conduction disorders)
  * Elevation of cardiac biomarkers (troponin)
  * Kinetic abnormalities on cardiac ultrasound
* Associated with ≥2 MRI criteria of tissue abnormality (edema, hyperhemia, myocardial fibrosis)
* Patient affiliated to a social security scheme or beneficiary of such a scheme
* No opposition to participation

Exclusion Criteria:

* Absence of documented coronary artery disease (cardiac CT or coronary angiography) or age <30 and low risk of coronary artery disease.
* Myocarditis secondary to immunotherapy.
* Presence of documented coronary artery disease (coronary angiography or cardiac CT)
* Presence of cardiomyopathy (hypertrophic cardiomyopathy, dilated cardiomyopathy)
* Infiltrative heart disease (sarcoidosis or cardiac amyloidosis)
* Severe valve disease
* Takotsubo
* Constrictive or chronic pericarditis
* Loeffler's endocarditis
* Non-compaction of the left ventricle
* Cardiac tumor
* Pulmonary embolism
* Coronary spasm
* Patients covered by articles L1121-5 to L1121-8 of the French Public Health Code (pregnant women, parturients, nursing mothers; persons deprived of liberty by judicial or administrative decision; protected adults)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient hospitalized for myocarditis at Grenoble Alpes University Hospital (CHUGA) or at Lyon University Hospital, with standardized reassessment at 3-6 months.
Sampling Method: Probability Sample
Enrollment: 244 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) rate at 4 years | 4 years
  MACE being defined by a composite criterion: 1) all-cause mortality, 2) cardiac decompensation requiring readmission, 3) cardiac transplantation,4) documented sustained ventricular arrhythmias >30s, 5) recurrence of myocarditis.

SECONDARY OUTCOMES:
Troponin us measured at 3 to 6 months | 3 to 6 months
  Prognostic value of troponin and MACE apparition. Troponin assays will be reported in ng/l.
  MACE being defined by a composite criterion: 1) all-cause mortality, 2) cardiac decompensation requiring readmission, 3) cardiac transplantation,4) documented sustained ventricular arrhythmias >30s, 5) recurrence of myocarditis. The MACE rate will be counted to answer the objective.
MACE apparition rate | 3 to 6 months
  Prognostic value of troponin and MACE apparition. Troponin assays will be reported in ng/l.
  MACE being defined by a composite criterion: 1) all-cause mortality, 2) cardiac decompensation requiring readmission, 3) cardiac transplantation,4) documented sustained ventricular arrhythmias >30s, 5) recurrence of myocarditis. The MACE rate will be counted to answer the objective.
Troponin us measured at 3 to 6 months | 3 to 6 months
  Prognostic value of Troponin us measured (in ng/l) at 3 to 6 months and watts generated on stress test at 3 to 6 months.
watts generated on stress test at 3 to 6 months | 3 to 6 months
  Prognostic value of Troponin us measured (in ng/l) at 3 to 6 months and watts generated on stress test at 3 to 6 months.
  Results of the stress test will be reported in watts.
Troponin Us measured at 3 to 6 months | 3 to 6 months
  Prognostic value of Troponin Us (ng/l) measured at 3 to 6 months and presence of abnormality on frequency holter Presence of abnormality on frequency holter is defined by the transition to atrial fibrillation and/or unsustained or sustained ventricular tachycardia.
Presence of abnormality on frequency holter (transition to atrial fibrillation and/or unsustained or sustained ventricular tachycardia). | 3 to 6 months
  Prognostic value of Troponin Us (ng/l) measured at 3 to 6 months and presence of abnormality on frequency holter Presence of abnormality on frequency holter is defined by the transition to atrial fibrillation and/or unsustained or sustained ventricular tachycardia.
  Presence of abnormality on frequency holter is defined by the transition to atrial fibrillation and/or unsustained or sustained ventricular tachycardia.
cardiac MRI. | 3 to 6 months
  Relationship between Troponin Us measured at 3 and 6 months and cardiac ultrasound measurements and cardiac MRI.
  Cardiac ultrasound measurements (longitudinal, radial and circumferential strain of the left ventricle in speckle tracking, left atrial strain in speckle tracking) Data collected during cardiac MRI are right and left ventricular function in percentage, cardiac mass in gram, and percentage of left ventricular fibrosis).
Troponin Us measured at 3 and 6 months | 3 to 6 months
  Relationship between Troponin Us measured at 3 and 6 months and cardiac ultrasound measurements and cardiac MRI.
  Cardiac ultrasound measurements (longitudinal, radial and circumferential strain of the left ventricle in speckle tracking, left atrial strain in speckle tracking) Data collected during cardiac MRI are right and left ventricular function in percentage, cardiac mass in gram, and percentage of left ventricular fibrosis).
cardiac ultrasound measurements | 3 to 6 months
  Relationship between Troponin Us measured at 3 and 6 months and cardiac ultrasound measurements and cardiac MRI.
  Cardiac ultrasound measurements (longitudinal, radial and circumferential strain of the left ventricle in speckle tracking, left atrial strain in speckle tracking) Data collected during cardiac MRI are right and left ventricular function in percentage, cardiac mass in gram, and percentage of left ventricular fibrosis).
The rate of occurrence of the following events at 30 days: ventricular arrhythmias, heart failure, need for heart transplantation, need for circulatory support, recovered cardiorespiratory arrest, all-cause mortality | 30 days
  Relationship between Troponin Us measured at 3 and 6 months and cardiac ultrasound measurements and cardiac MRI.
  Cardiac ultrasound measurements (longitudinal, radial and circumferential strain of the left ventricle in speckle tracking, left atrial strain in speckle tracking) Data collected during cardiac MRI are right and left ventricular function in percentage, cardiac mass in gram, and percentage of left ventricular fibrosis).

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble University Hospital, La Tronche, France

REFERENCES:
- [Background] Ammirati E, Frigerio M, Adler ED, Basso C, Birnie DH, Brambatti M, Friedrich MG, Klingel K, Lehtonen J, Moslehi JJ, Pedrotti P, Rimoldi OE, Schultheiss HP, Tschope C, Cooper LT Jr, Camici PG. Management of Acute Myocarditis and Chronic Inflammatory Cardiomyopathy: An Expert Consensus Document. Circ Heart Fail. 2020 Nov;13(11):e007405. doi: 10.1161/CIRCHEARTFAILURE.120.007405. Epub 2020 Nov 12. PMID 33176455
- [Background] Caforio AL, Pankuweit S, Arbustini E, Basso C, Gimeno-Blanes J, Felix SB, Fu M, Helio T, Heymans S, Jahns R, Klingel K, Linhart A, Maisch B, McKenna W, Mogensen J, Pinto YM, Ristic A, Schultheiss HP, Seggewiss H, Tavazzi L, Thiene G, Yilmaz A, Charron P, Elliott PM; European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Current state of knowledge on aetiology, diagnosis, management, and therapy of myocarditis: a position statement of the European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Eur Heart J. 2013 Sep;34(33):2636-48, 2648a-2648d. doi: 10.1093/eurheartj/eht210. Epub 2013 Jul 3. PMID 23824828
- [Background] Barone-Rochette G, Augier C, Rodiere M, Quesada JL, Foote A, Bouvaist H, Marliere S, Fagret D, Baguet JP, Vanzetto G. Potentially simple score of late gadolinium enhancement cardiac MR in acute myocarditis outcome. J Magn Reson Imaging. 2014 Dec;40(6):1347-54. doi: 10.1002/jmri.24504. Epub 2013 Dec 1. PMID 24293405
- [Background] Dedic A, Lubbers MM, Schaap J, Lammers J, Lamfers EJ, Rensing BJ, Braam RL, Nathoe HM, Post JC, Nielen T, Beelen D, le Cocq d'Armandville MC, Rood PP, Schultz CJ, Moelker A, Ouhlous M, Boersma E, Nieman K. Coronary CT Angiography for Suspected ACS in the Era of High-Sensitivity Troponins: Randomized Multicenter Study. J Am Coll Cardiol. 2016 Jan 5;67(1):16-26. doi: 10.1016/j.jacc.2015.10.045. PMID 26764061
- [Background] Aquaro GD, Perfetti M, Camastra G, Monti L, Dellegrottaglie S, Moro C, Pepe A, Todiere G, Lanzillo C, Scatteia A, Di Roma M, Pontone G, Perazzolo Marra M, Barison A, Di Bella G; Cardiac Magnetic Resonance Working Group of the Italian Society of Cardiology. Cardiac MR With Late Gadolinium Enhancement in Acute Myocarditis With Preserved Systolic Function: ITAMY Study. J Am Coll Cardiol. 2017 Oct 17;70(16):1977-1987. doi: 10.1016/j.jacc.2017.08.044. PMID 29025554
- [Background] Grani C, Eichhorn C, Biere L, Murthy VL, Agarwal V, Kaneko K, Cuddy S, Aghayev A, Steigner M, Blankstein R, Jerosch-Herold M, Kwong RY. Prognostic Value of Cardiac Magnetic Resonance Tissue Characterization in Risk Stratifying Patients With Suspected Myocarditis. J Am Coll Cardiol. 2017 Oct 17;70(16):1964-1976. doi: 10.1016/j.jacc.2017.08.050. PMID 29025553
- [Background] Wong BTW, Christiansen JP. Clinical Characteristics and Prognostic Factors of Myocarditis in New Zealand Patients. Heart Lung Circ. 2020 Aug;29(8):1139-1145. doi: 10.1016/j.hlc.2020.01.007. Epub 2020 Feb 17. PMID 32094080